CLINICAL TRIAL: NCT06614517
Title: EVALUATION OF BIRD WATCHING IN REDUCING STRESS AMONG UNIVERSITY STUDENTS
Brief Title: Bird Watching to Reduce Stress in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Principal Investigator, Leidy Johanna Rueda Díaz, Associate Professor, Universidad Industrial de Santander
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4217
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-03

CONDITIONS: Stress, Psychologic
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Birdwatching Intervention Arm (Experimental): The intervention arm will involve participants, divided into four subgroups, taking part in field trips for visual and auditory birdwatching. These trips will take place every 15 days over three sessions, guided by an expert in the subject. Students will be provided with binoculars and guidance on the use of apps to identify observed birds. Additionally, WhatsApp groups will be created for each subgroup, where videos and audios of birds will be shared, along with weekly challenges to reinforce exposure to the intervention. The outings will take place in natural environments such as coffee farms and forests near Bucaramanga.
  Interventions: Other: Birdwatching Intervention
- Control Arm (No Intervention): The control group will not receive any intervention related to birdwatching. Participants in this group will continue with their usual activities without taking part in the field trips or complementary activities such as watching videos or listening to bird sounds.

INTERVENTIONS:
Other: Birdwatching Intervention — Description: Participants will attend three birdwatching sessions, where they will enjoy direct contact with nature in selected environments such as forests and farms. These outings will be guided by an expert, who will also introduce participants to the use of binoculars and tools for identifying the birds observed during the excursions. During the outings, participants will learn the body scan technique, which will help them focus on physical sensations without making judgments. This exercise will encourage them to pay attention to details such as muscle tension, temperature, or surface contact, allowing them to be more present and connected to their surroundings during the birdwatching sessions. In addition to the in-person outings, participants will receive digital materials via WhatsApp to complement the intervention.Birdwatching Intervention
  Arms: Birdwatching Intervention Arm

SUMMARY:
The goal of this study is to learn if birdwatching can reduce stress in university students. It will also explore students; experiences with the intervention. The main questions it aims to answer are:

Does birdwatching reduce students perceived stress levels? What are the experiences of students who participate in the birdwatching intervention? Why do some students drop out of the study? Researchers will compare a group of students who participate in birdwatching outings to a control group that does not receive the intervention to determine if birdwatching is effective in reducing stress.

Participants will:

Either participate in birdwatching outings or be in a control group with no intervention Complete a perceived stress scale (PSS-10) to measure their stress levels Take part in semi-structured interviews to discuss their experiences with the intervention or their reasons for dropping out of the study

ELIGIBILITY:
Inclusion Criteria:

* University students who meet the following inclusion criteria will be included in the study: being 18 years of age or older, being enrolled in any undergraduate program at the Universidad Industrial de Santander, having a score of 10 or higher on the Perceived Stress Scale (PSS-10), and having access to WhatsApp.

Exclusion Criteria:

* University students with a medical diagnosis of any mental illness under pharmacological or non-pharmacological treatment, with health conditions that prevent them from seeing, hearing, or moving, as well as students who have engaged in birdwatching in the last six months, will not be included.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Adherence to the intervention | From enrollment to the three follow-up evaluations at 6, 9, and 17 weeks after assignment to the intervention or control group
  To determine adherence to the intervention, the proportion of students who successfully completed the number of sessions and challenges outlined in the intervention protocol will be calculated, as well as the number of university students who dropped out of the intervention
The Perceived Stress Scale | From enrollment to the three follow-up evaluations at 6, 9, and 17 weeks after assignment to the intervention or control group.
  Perceived Stress Scale: (PSS-10). This instrument measures the level of perceived stress during the last month. It consists of 10 questions with a five-option Likert-type response format. The score ranges from 0 to 40. A higher score indicates a higher level of perceived stress.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Scale (GAD-7) | From enrollment to the three follow-up evaluations at 6, 9, and 17 weeks after assignment to the intervention or control group
  The GAD-7 is used to measure anxiety symptoms. It consists of 7 items, each rated on a scale from 0 to 3, with total scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptoms.
Patient Health Questionnaire (PHQ-9) | From enrollment to the three follow-up evaluations at 6, 9, and 17 weeks after assignment to the intervention or control group
  The PHQ-9 is a self-report outcome questionnaire used to screen for depressive symptoms. It consists of 9 items. Responses are scored on a scale from 0 to 3, with total scores ranging from 0 to 27. Higher scores indicate more severe depression.
Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the three follow-up evaluations at 6, 9, and 17 weeks after assignment to the intervention or control group
  It consists of 19 self-administered questions, rated on a scale from 0 to 3, generating an overall score from 0 to 21. Higher overall scores represent worse subjective sleep quality.

OTHER OUTCOMES:
Feasibility- implementation of the intervention | From inclusion in the study until the last follow up at 17 weeks
  The Feasibility of Intervention measure gauges how practical and possible it is to implement an intervention within a given setting. Semi-structured interviews with the interveners.
Feasibility - Enrollment | From the first day of study recruitment until the date of the last participant to complete the intervention, assessed up to 17 weeks
  Enrollment rates calculated as percentage of enrolled vs interested participants
Experiance | From inclusion in the study until the last follow up at 17 weeks
  Semi-structured interviews with study participants.
Participant Attrition Rate | Up to 17 weeks after study start
  Percentage of enrolled participants who withdraw or are lost to follow-up before completion of study procedures. Unit of Measure: Percentage.
Overall compliance | From day of recruitment of the first participant to day of the last follow-up meeting of the last participant, assessed up to 17 weeks.
  Number of participants that completed all questionnaires at baseline, 6 weeks, 9 weeks and 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: LEIDY J RUEDA DÍAZ, PhD, Principal Investigator — Universidad Industrial de Santander
Locations (1):
- Universidad Industrial de Santander, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication